CLINICAL TRIAL: NCT05198674
Title: The SPYRAL AFFIRM Global Clinical Study of Renal Denervation With the Symplicity Spyral Renal Denervation System in Subjects With Uncontrolled Hypertension (SPYRAL AFFIRM)
Brief Title: SPYRAL AFFIRM Global Study of RDN With the Symplicity Spyral RDN System in Subjects With Uncontrolled HTN
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Vascular (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MDT20044RDN004; SPYRAL SWFYT (NCT07115953) (Other: ClinicalTrials.gov)
Record Dates: First submitted 2021-11-05; First posted 2022-01-20 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-09

CONDITIONS: Hypertension; Vascular Diseases; Cardiovascular Diseases; Chronic Kidney Diseases; Diabetes Mellitus
MeSH Terms: conditions — Hypertension; Vascular Diseases; Cardiovascular Diseases; Renal Insufficiency, Chronic; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Main Cohort: Renal Denervation (Experimental): Renal angiography and Renal Denervation (Symplicity Spyral™ multi-electrode renal denervation system)
  Interventions: Device: Renal Denervation (Symplicity Spyral™)

INTERVENTIONS:
Device: Renal Denervation (Symplicity Spyral™) — Device: Symplicity Spyral™ multi-electrode renal denervation system. After a renal angiography according to standard procedures, subjects are treated with the renal denervation procedure.
  Other Names: Renal Angiography; Renal Denervation

SUMMARY:
The purpose of this single-arm interventional study is to evaluate the long-term safety, efficacy, and durability of the Symplicity Spyral system in subjects treated with renal denervation.

Additionally, long-term follow-up data will also be collected from eligible subjects previously treated in the SPYRAL PIVOTAL-SPYRAL HTN-OFF MED and SPYRAL HTN-ON MED studies.

ELIGIBILITY:
Inclusion Criteria:

1. Individual is diagnosed with hypertension and has a baseline office systolic blood pressure ≥140 mmHg
2. Individual has a baseline office diastolic blood pressure ≥ 90 mmHg
3. Individual has an average systolic baseline home blood pressure ≥135 mmHg

Exclusion Criteria:

1. Individual lacks appropriate renal artery anatomy
2. Individual has undergone prior renal denervation
3. Individual has a documented condition that would prohibit or interfere with ability to obtain an accurate blood pressure measurement
4. Individual requires chronic oxygen support or mechanical ventilation other than nocturnal respiratory support for sleep apnea
5. Individual has an estimated glomerular filtration rate (eGFR) of <45
6. Individual has one or more episode(s) of orthostatic hypotension
7. Individual is pregnant, nursing or planning to become pregnant
8. Individual has primary pulmonary hypertension
9. Individual has documented type 1 diabetes mellitus or poorly-controlled type 2 diabetes mellitus with glycosylated hemoglobin greater than 8.0%

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1300 (Estimated)
Dates: Start 2021-10-20 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2029-11-30 (Estimated)

PRIMARY OUTCOMES:
The Primary endpoint of office Systolic Blood Pressure (SBP) change at 6 months. | 6 months
  The Primary endpoint of office Systolic Blood Pressure (SBP) change at 6 months will be assessed for all patients in the Main Study Cohort

SECONDARY OUTCOMES:
Office Systolic Blood Pressure change | From baseline to 3, 6, 12, 24, and 36 months post-procedure
Home Blood Pressure change (Main Cohort Only) | From baseline to 3, 6, 12, 24, and 36 months post-procedure
Change in blood pressure as measured by 24-hour ABPM | From baseline to 3, 6, 12, 24, and 36 months post-procedure
Percent of subjects achieving blood pressure control as measured by OBP, HBP and ABPM | From baseline to 3, 6, 12, 24, and 36 months post-procedure
Time subject's blood pressure is controlled | Procedure to 36 months post-procedure
Change in number of anti-hypertensive medications taken from baseline | From baseline to 3, 6, 12, 24, and 36 months post-procedure
Change from baseline in EQ-5D quality of life score | From baseline to 3, 6, 12, 24, and 36 months post-procedure
Change from baseline in hypertension health status score | From baseline to 3, 6, 12, 24, and 36 months post-procedure
Evaluate pre-specified subgroups (Chronic Kidney Disease, Diabetes Mellitus Type II, etc) as predictors for change in blood pressure as measured by OBP, HBP and ABPM | From baseline to 3, 6, 12, 24, and 36 months post-procedure
Evaluation of slope of eGFR | From baseline to 3, 6, 12, 24, and 36 months post-procedure
Incidence of events, including major adverse events | From baseline to 3, 6, 12, 24, and 36 months post-procedure

CONTACTS AND LOCATIONS:
Overall Officials: David Kandzari, MD, Principal Investigator — Piedmont Heart Institute; Felix Mahfoud, MD, Principal Investigator — Saarland University Hospital
Locations (100):
- United States (79):
  - University of Alabama at Birmingham (UAB) Hospital, Birmingham, Alabama
  - Banner Heart Hospital, Mesa, Arizona
  - Abrazo Arizona Heart Hospital/Biltmore Cardiology, Phoenix, Arizona
  - HonorHealth Research Institute, Scottsdale, Arizona
  - Arkansas Cardiology, Little Rock, Arkansas
  - Scripps Memorial Hospital, La Jolla, California
  - University of California, San Francisco, San Francisco, California
  - Stanford Hospital and Clinics, Stanford, California
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - Colorado Heart and Vascular PC, Lakewood, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - BayCare Health System, Clearwater, Florida
  - Clearwater Cardiovascular Consultants, Clearwater, Florida
  - Baptist Medical Center, Jacksonville, Florida
  - University of Miami Hosptial, Miami, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Orlando Health Heart & Vascular Institute, Orlando, Florida
  - BayCare Medical Group, Safety Harbor, Florida
  - Tallahassee Memorial Healthcare, Inc, Tallahassee, Florida
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Piedmont Heart Institute, Atlanta, Georgia
  - Wellstar Research Institute, Marietta, Georgia
  - University of Chicago Medicine, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Heart Care Centers of Illinois, Palos Park, Illinois
  - St. Vincents Hospital, Indianapolis, Indiana
  - Mercy Medical Center, West Des Moines, Iowa
  - The Johns Hopkins Hospital, Baltimore, Maryland
  - Saint Joseph Medical Center (Towson MD), Towson, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Henry Ford Saint John Hospital, Detroit, Michigan
  - Spectrum Health Hospitals, Grand Rapids, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Henry Ford Providence Southfield Hospital, Southfield, Michigan
  - Metropolitan Heart and Vascular Institute (MHVI), Coon Rapids, Minnesota
  - CentraCare Heart & Vascular Center, Saint Cloud, Minnesota
  - North Mississippi Medical Center, Tupelo, Mississippi
  - University of Nebraska Medical Center, Omaha, Nebraska
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Dartmouth-Hitchcock, Lebanon, New Hampshire
  - Virtua Medical Group, Marlton, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Jersey Shore University Medical Center, Neptune City, New Jersey
  - The Valley Hospital, Paramus, New Jersey
  - SJH Cardiology Associates, Liverpool, New York
  - North Shore University Hospital, Manhasset, New York
  - Weill Cornell Medical Center, New York, New York
  - Saint Francis Hospital, Roslyn, New York
  - Montefiore Medical Center, The Bronx, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Sanford Medical Center, Fargo, North Dakota
  - The Lindner Center, Cincinnati, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Cleveland Cl inic, Cleveland, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Oklahoma Heart Hospital, Oklahoma City, Oklahoma
  - UPMC Harrisburg Hospital, Harrisburg, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Rhode Island Hospital and Health Services, Providence, Rhode Island
  - AnMed Health Medical Center, Anderson, South Carolina
  - Centennial Medical Center, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor Jack and Jane Hamilton Heart and Vascular Hospital, Dallas, Texas
  - DHR Health Institute for Research and Development, Edinburg, Texas
  - Houston Methodist, Houston, Texas
  - Baylor Scott & White The Heart Hospital Baylor Plano, Plano, Texas
  - Methodist Hospital, San Antonio, Texas
  - The University of Texas at Tyler, Tyler, Texas
  - Intermountain Medical Center, Murray, Utah
  - University of Vermont Medical Center, Burlington, Vermont
  - UVA Medical Center, Charlottesville, Virginia
  - Providence Regional Medical Center Everett, Everett, Washington
  - West Virginia University, Morgantown, West Virginia
  - Advocate Aurora Health-Aurora St. Luke's Medical Center (ASLMC), Milwaukee, Wisconsin
- Australia (2):
  - The Alfred Hospital, Melbourne, Victoria
  - Royal Perth Hospital (Dobney Hypertension Centre), Perth, Western Australia
- Belgium (5):
  - Algemeen Stedelijk Ziekenhuis - R&D Hartziekten, Aalst, Oost - Vlaanderen
  - AZ Sint Jan Brugge-Oostende av, Bruges
  - Ziekenhuis Oost Limburg - Campus Sint-Jan, Genk
  - University Hospital Ghent, Ghent
  - Chc Montlegia, Liège
- France (2):
  - Hôpital Saint André -Centre Hospitalier Universitaire de Bordeaux, Bordeaux
  - Hôpital Pitié Salpêtrière, Paris
- Germany (5):
  - Uniklinik Erlangen, Erlangen
  - Justus-Liebig-Universität Gießen, Giessen
  - Universitatsklinikum des Saarlandes, Homburg
  - Herzzentrum Leipzig, Leipzig
  - Sana Kliniken Lübeck GmbH, Lübeck
- Hippokration General Hospital of Athens, Athens, Greece
- Mater Misericordiae University Hospital, Dublin, Dublin, Ireland
- Centre Hospitalier Princesse Grace, Monaco, Monaco
- Netherlands (2):
  - Zuyderland Medisch Centrum Heerlen, Heerlen
  - Erasmus Universtiy Medical Center, Rotterdam
- Danderyd Sjukhus, Stockholm, Sweden
- John Radcliffe Hospital, Oxford, Oxfordshire, United Kingdom

REFERENCES:
- [Derived] Abid S, Mehta S, Munazzah F, Yager N, Baloch S, Hongalgi K. Renal Denervation: A New Era in the Management of Resistant Hypertension. Kidney360. 2025 Nov 1;6(11):2010-2016. doi: 10.34067/KID.0000000961. Epub 2025 Aug 13. PMID 40802676